CLINICAL TRIAL: NCT07149038
Title: A Single-Center, Randomized, Double-Blind Feasibility Trial Assessing the Initial Efficacy and Safety of Cerogrin, a Medical Device for Auricular Vagus Nerve Stimulation, in Improving Cognition in Patients With Vascular Dementia or Vascular Mild Cognitive Impairment: A Comparison With Sham Control
Brief Title: Evaluation of Cerogrin for Auricular Vagus Nerve Stimulation in Vascular Dementia or Vascular Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurogrin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NG-VCI-01
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Vascular Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia, Vascular; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerogrin Group (Experimental): Participants in this group will receive transcutaneous auricular vagus nerve stimulation using the Cerogrin device.
  Interventions: Device: Cerogrin
- Sham Group (Sham Comparator): Participants in this group will use a sham device identical in appearance to the Cerogrin device but delivering no stimulation.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Cerogrin — Participants in this arm will receive transcutaneous auricular vagus nerve stimulation using the Cerogrin device. This device non-invasively delivers electrical stimulation to the vagus nerve located on the outer ear, aiming to improve cognitive function.
  Arms: Cerogrin Group
Device: Sham Device — Participants in this arm will use a sham device. This device is identical in appearance to the active Cerogrin device but delivers no electrical stimulation or therapeutic effect. The sham device serves as a control to compare outcomes with the active treatment group.
  Arms: Sham Group

SUMMARY:
This clinical trial evaluates the preliminary effectiveness and safety of Cerogrin, a medical device developed by Neurogrin Inc. for auricular vagus nerve stimulation, in patients with vascular dementia or vascular mild cognitive impairment. Given the limited availability of effective pharmacological treatments for these conditions, the study aims to assess whether Cerogrin can enhance cognitive function through non-invasive neuromodulation.

Twenty-four participants will be randomized to receive either the active Cerogrin device or a sham (non-stimulating) device. Daily use will occur at home for 30 minutes over a four-week intervention period. The full study duration, including baseline assessments and follow-up, will span up to three months. During this period, cognitive function, neural activity, and safety outcomes will be systematically evaluated. This feasibility trial represents a critical step toward expanding therapeutic options for vascular cognitive impairment.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 55 to 89 years.
* Diagnosed with vascular dementia or vascular mild cognitive impairment within 1 year before screening, with subcortical lesions confirmed on MRI.
* For both diagnoses:
* Severe white matter hyperintensity on MRI (Fazekas scale: deep white matter ≥ 2.5 cm or caps/bands ≥ 1.0 cm).
* Z-score < -1.0 SD in at least one cognitive domain (adjusted for education, age, and sex).
* For vascular dementia: independence in daily living impaired.
* For vascular mild cognitive impairment: independence in daily living preserved.
* K-MMSE-II score ≥ 18 and CDR score 0.5 to 1.0 at screening.
* Stable cognitive-enhancing medication (if applicable) for ≥4 weeks before baseline.
* Availability of a caregiver (at least 8 hours/week contact).
* Females of childbearing potential: agreement to use medically acceptable contraception during the study.
* Provided written informed consent.
* Willingness to comply with study protocol.

Exclusion Criteria

* Dementia other than vascular dementia (e.g., Alzheimer's disease, Lewy body dementia, frontotemporal dementia).
* Conditions causing cognitive decline (e.g., uncontrolled metabolic diseases, CNS infections, cerebrovascular disease, traumatic brain injury, Parkinson's disease).
* Severe psychiatric disorders (e.g., major depression, schizophrenia, substance abuse).
* Serious unstable physical conditions.
* MRI contraindications (e.g., claustrophobia, metal implants, contrast agent allergy).
* Auricular skin disease or condition preventing device use.
* Inability to comply with study procedures.
* Pregnancy or breastfeeding.
* Participation in other clinical trials within 30 days before screening.
* Any other condition deemed inappropriate for participation by the investigator.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  The CDR-SB is a scale that evaluates a patient's cognitive function and ability to live independently. The scores range from 0 to 18, with higher scores indicating more severe cognitive impairment.
Change from Baseline in Korean Montreal Cognitive Assessment (K-MoCA) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  he K-MoCA is a cognitive screening tool used to detect mild cognitive impairment. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Change from Baseline in Korean Mini-Mental State Examination-2 (K-MMSE-II) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  The K-MMSE-II is a cognitive screening test used to assess a person's cognitive function, with scores ranging from 0 to 30.
Change from Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-cog 13) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  The ADAS-cog 13 is a scale used to assess the severity of cognitive symptoms in Alzheimer's disease. Higher scores indicate greater cognitive impairment.
Change from Baseline in Controlled Oral Word Association Test (COWAT) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  This test measures a person's verbal fluency and executive function.
Change from Baseline in Stroop Test Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  The Stroop test measures a person's cognitive flexibility and executive function.
Change from Baseline in Trail Making Test (TMT) Score | Baseline to Week 4 (End of Intervention Period) and/or Week 8 (End of Follow-up)
  The TMT is a neuro-psychological test of visual attention and task switching.

SECONDARY OUTCOMES:
Change from Baseline in DTI-ALPS Score on Magnetic Resonance Imaging (MRI) | Baseline to Week 4 (End of Intervention Period)
  This score evaluates the brain's perivascular space, which is related to cerebral small vessel disease.
Change from Baseline in Brain Function using Functional Magnetic Resonance Imaging (fMRI) | Baseline to Week 4 (End of Intervention Period)
  This method measures brain activity by detecting changes in blood flow.
Change from Baseline in Electroencephalogram (EEG) Brain Wave Analysis | Baseline to Week 4 (End of Intervention Period)
  Descriptive statistics (number of subjects, mean, standard deviation, median, minimum, and maximum) for changes in EEG power and relative EEG power by brainwave frequency band will be presented for each group. Statistical significance of the differences between groups will be tested using ANCOVA, with the indication (vascular dementia/vascular mild cognitive impairment) and baseline relative EEG power as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Jaeho Kim, M.D., Ph.D., Principal Investigator — Hallym University Dongtan Sacred Heart Hospital
Locations (1):
- Dongtan Hallym University Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No